CLINICAL TRIAL: NCT03637959
Title: Liver Fibrosis Evaluation Using Ultrasound Shear Wave Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shiago Chen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-002289; R01DK106957 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mechanical Vibrations with Ultrasound Shear Wave Imaging (Experimental): Subjects that are scheduled to undergo a clinical indicated Magnetic Resonance Elastography (MRE) will also have mechanical vibrations ultrasound shear wave imaging to measure liver stiffness
  Interventions: Device: Mechanical Vibrations with Ultrasound Shear Wave Imaging

INTERVENTIONS:
Device: Mechanical Vibrations with Ultrasound Shear Wave Imaging — Multiple miniature mechanical vibrators will be placed on the body surface of rib cage of the subject or introduced through an audio loudspeaker in contact with the subject's upper torso or through miniature vibrator attached to the ultrasound probe. Repeated ultrasound stiffness measurements will be made at different locations within the liver parenchyma while the mini vibrators introduce shear wave in the liver, similar to an MRE examination.

SUMMARY:
The Researchers are trying to assess the effectiveness of a new ultrasound technique for non-invasive evaluation of liver fibrosis.

DETAILED DESCRIPTION:
Utilizing vibrating transducer, receiver and speaker in differing sequences, while collecting ultrasound liver tissue elastography measurements during participant breath holds. Participants fast for a minimum of four hours and are positioned lying on left side with knees slightly bent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers or patients who are scheduled for clinically indicated liver MRE for fibrosis staging.
* Age 18 to 80.

Exclusion Criteria:

* Subjects lacking capacity to consent
* Subjects with unreliable ultrasound or MRE measurements.
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigao Chen, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mechanical Vibrations With Ultrasound Shear Wave Imaging
Started | 270
Completed | 270
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mechanical Vibrations With Ultrasound Shear Wave Imaging
Number analyzed (Participants) | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 256
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 250
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 270

OUTCOME MEASURES:

1. Primary Outcome: Liver Stiffness Measured by MRE
Description: Liver stiffness measured by standard of care Magnetic Resonance Elastography reported in Kilopascals (kPa) (used as a benchmark reference in this study).
Time Frame: Baseline, approximately 1 day
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Mechanical Vibrations With Ultrasound Shear Wave Imaging
Number analyzed (Participants) | 270
kPa | 3.07 (1.36)

2. Primary Outcome: Liver Stiffness Measured by Mechanical Vibrations With Ultrasound Shear Wave Imaging
Description: Liver stiffness measured by Mechanical Vibrations with Ultrasound Shear Wave Imaging reported in kilopascal (kPa).
Time Frame: Baseline, approximately 1 day
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Mechanical Vibrations With Ultrasound Shear Wave Imaging
Number analyzed (Participants) | 270
kPa | 2.66 (1.00)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to completion of study imaging for a total of approximately 1 day on all participants.
Arm/Group | Mechanical Vibrations With Ultrasound Shear Wave Imaging
All-Cause Mortality (participants affected / at risk) | 0/270
Serious Adverse Events (participants affected / at risk) | 0/270
Other Adverse Events (participants affected / at risk) | 0/270

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT03637959/Prot_SAP_002.pdf